CLINICAL TRIAL: NCT02027467
Title: Assessment of the Effect of StemAlive® Herbal Supplement on the Levels of Circulating Hematopoietic Stem Cells in Human Volunteers
Brief Title: Study to Assess the Effect of StemAlive® Supplement on the Levels of Stem Cells in Human Volunteers
Acronym: Hematoalive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Stem Vida International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SV/121108/SA/HSC
Record Dates: First submitted 2013-11-18; First posted 2014-01-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Hematopoietic stem cells; Herbal; Dietary; CD cells; Basic research

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- StemAlive® (Experimental): Stem Alive® includes ingredients like green tea, ashwagandha. Dose: 3 capsules twice daily to be taken orally for 14 days.
  Interventions: Dietary Supplement: StemAlive®
- Placebo (Placebo Comparator): Matching placebo capsules (for StemAlive®) containing polyethylene glycol, rice powder and magnesium stearate. Dose: 3 capsules twice daily to be taken orally for 14 days.
  Interventions: Dietary Supplement: Placebo (For StemAlive®)

INTERVENTIONS:
Dietary Supplement: StemAlive®
  Arms: StemAlive®
Dietary Supplement: Placebo (For StemAlive®)
  Arms: Placebo

SUMMARY:
Combination of various herbs is known to promote mobilization of hematopoietic stem cells. Hence the current study has been intended to study the effect of Stem Alive® on mobilization of stem cells. Stem Alive® include ingredients like green tea, ashwagandha, etc which are known to be used as traditional medicine. They are also tested qualitatively in academic and nutritional science research centers throughout the world and which substantially according to those studies stimulate the augmented availability of circulating hematopoietic cells. This study is projected to investigate the mobilization of stem cells on healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male and Female Volunteers
* Willing to sign Informed Consent Form

Exclusion Criteria:

* Anemia
* SGOT and Serum Creatinine values twice the upper limit of normal
* Volunteers who smoke / consume alcohol / take recreational drugs
* Fever or Flu in the last one week of screening
* History of Gastric or Duodenal Ulcer
* Volunteers on vitamins, nutritional or herbal products since last one month
* Pregnant, Breast feeding and Lactating women
* Volunteers taking antibiotic, NSAIDS, anti-inflammatory within last 7 days
* Allergic to ingredients of test product
* Any co morbid or systemic condition or immunocompromised state making volunteer unfit for participation.
* Volunteers deemed unfit for the study by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
CD34+ | Day 0, Day 1, Day 2, Day 7, Day 12 and Day 14
CD45+ | Day 0, Day 1, Day 2, Day 7, Day 12 and Day 14
CD133+ | Day 0, Day 1, Day 2, Day 7, Day 12 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Patil, MD, Principal Investigator
Locations (1):
- Dhanwantari Clinic, Mumbai, Maharashtra, India